CLINICAL TRIAL: NCT06543576
Title: A Prospective Cohort Study of Integrating Radiotherapy Into Chemotherapy With Pembrolizumab and Bevacizumab in Newly Diagnosed Stage IVB Cervical Cancer
Brief Title: External Beam Radiation Therapy and Brachytherapy With Chemotherapy and Immunotherapy for the Treatment of Stage IVB Cervical Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-000095; NCI-2024-06183 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-000095 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-05

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Squamous Cell Carcinoma; Stage IVB Cervical Cancer American Joint Committee on Cancer (AJCC) v8
MeSH Terms: interventions — Bevacizumab; Immunoglobulin G; Disulfides; Specimen Handling; Brachytherapy; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Congresses as Topic; Radiation; Paclitaxel; Taxes; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (EBRT, brachytherapy, chemotherapy, immunotherapy) (Experimental): PART 1: Patients receive cisplatin IV, paclitaxel IV, pembrolizumab IV over 30 minutes, and bevacizumab IV on day 1 of each cycle. Cycles repeat every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients receive no treatment for 3 weeks.
  PART 2: Patients undergo EBRT for 25 treatments delivered over 5 weeks, and brachytherapy over 3-5 treatments. Patients also receive pembrolizumab IV over 30 minutes and bevacizumab IV on day 1 of each cycle. Cycles for immunotherapy repeat every 21 days for a total of 2 years in the absence of disease progression or unacceptable toxicity. Participants who complete study intervention after 2 years of pembrolizumab are eligible for up to 1 year of additional pembrolizumab (second course) upon experiencing disease progression.
  Patients undergo CT, PET/CT, and/or MRI throughout the study. Patients also undergo blood sample collection throughout the study.
  Interventions: Biological: Bevacizumab; Procedure: Biospecimen Collection; Radiation: Brachytherapy; Drug: Cisplatin; Radiation: External Beam Radiation Therapy; Drug: Paclitaxel; Biological: Pembrolizumab; Other: Questionnaire Administration

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Mvasi; MYL-1402O; Onbevzi; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Radiation: Brachytherapy — Undergo brachytherapy
  Other Names: Brachytherapy, NOS; Internal Radiation; Internal Radiation Brachytherapy; Internal Radiation Therapy; Radiation Brachytherapy; Radiation, Internal
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam Radiotherapy (conventional); External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; QL2107; SCH 900475; SCH-900475; SCH900475
Other: Questionnaire Administration — Ancillary study

SUMMARY:
This phase I/II trial tests the safety and effectiveness of receiving external beam radiation therapy (EBRT) and brachytherapy along with chemotherapy, consisting of cisplatin and paclitaxel, and immunotherapy, consisting of bevacizumab and pembrolizumab, for the treatment of patients with stage IVB cervical cancer. EBRT is type of radiation therapy that uses a machine to aim high-energy rays at the cancer from outside of the body. Brachytherapy, also known as internal radiation therapy, uses radioactive material placed directly into or near a tumor to kill tumor cells. Cisplatin is in a class of medications known as platinum-containing compounds. It works by killing, stopping or slowing the growth of tumor cells. Paclitaxel is in a class of medications called antimicrotubule agents. It stops tumor cells from growing and dividing and may kill them. Bevacizumab is in a class of medications called antiangiogenic agents. It works by stopping the formation of blood vessels that bring oxygen and nutrients to tumor. This may slow the growth and spread of tumor. A monoclonal antibody, such as pembrolizumab, is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Giving EBRT and brachytherapy along with chemotherapy and immunotherapy may be a safe and effective way to treat patients with stage IVB cervical cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate that radiotherapy can be safely integrated into chemotherapy and pembrolizumab with bevacizumab in newly diagnosed stage IVB cervical cancer to improve outcomes.

SECONDARY OBJECTIVE:

I. To demonstrate improvements with overall response rate, overall survival (OS), and duration of response with the addition of radiation therapy to standard of care in stage IVB cervical cancer.

EXPLORATORY OBJECTIVES:

I. To demonstrate improved quality of life and disease-related toxicity with the addition of radiation therapy to standard of care chemotherapy in stage IVB cervical cancer.

II. To explore the association of known risk factors (age, race/ethnicity, smoking status, baseline quality of life, combined positive score [CPS] score 1-10 versus > 10, and performance status with the change in QOL, treatment outcomes, and toxicities.

III. To explore circulating tumor deoxyribonucleic acid (ctDNA) as a biomarker to monitor the response to upfront chemotherapy-immunotherapy and subsequent radiation.

IV. To use T cell receptor repertoire sequencing (TCRseq) to define T cell clones present in the tumor and to establish their concordance with peripheral blood T cell clones at baseline and in response to therapy.

OUTLINE:

PART 1: Patients receive cisplatin intravenously (IV), paclitaxel IV, pembrolizumab IV over 30 minutes, and bevacizumab IV on day 1 of each cycle. Cycles repeat every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients receive no treatment for 3 weeks.

PART 2: Patients undergo EBRT for 25 treatments delivered over 5 weeks, and brachytherapy over 3-5 treatments. Patients also receive pembrolizumab IV over 30 minutes and bevacizumab IV on day 1 of each cycle. Cycles for immunotherapy repeat every 21 days for a total of 2 years in the absence of disease progression or unacceptable toxicity. Participants who complete study intervention after 2 years of pembrolizumab are eligible for up to 1 year of additional pembrolizumab (second course) upon experiencing disease progression.

Patients undergo computed tomography (CT), positron emission tomography (PET)/CT, and/or magnetic resonance imaging (MRI) throughout the study. Patients also undergo blood sample collection throughout the study.

After completion of study treatment, patients follow up at 30 days and every 6 weeks for up to 1 year then every 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of Stage IVB cervical cancer will be enrolled in this study
* Patients with stage IVB adenocarcinoma, adenosquamous carcinoma, or squamous-cell carcinoma of the cervix that has not yet been treated with systemic chemotherapy or radiation therapy
* Participants who have adverse events (AEs) due to previous anticancer therapies must have recovered to ≤ grade 1 or baseline. Participants with endocrine-related AEs who are adequately treated with hormone replacement or participants who have ≤ grade 2 neuropathy are eligible
* The participant provides written informed consent for the trial
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
* Archival tumor tissue sample or newly obtained [core, incisional or excisional] biopsy of a tumor lesion not previously irradiated has been provided. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue
* Patients must have PD-L1 status, CPS score of over 1. PD-L1 status will be determined per institutional standards via the Food and Drug Administration (FDA)-approved test, Dako PD-L1 immunohistochemistry (IHC) 22C3 pharmDx kit with combined positive score (CPS) interpretation
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) anti-viral therapy for at least 4 weeks, and have undetectable HBV viral load prior to randomization.

Note: Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.

Hepatitis B screening tests are not required unless:

* Known history of HBV infection
* As mandated by local health authority

  * Participants with a history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening.

Note: Participants must have completed curative anti-viral therapy at least 4 weeks prior to randomization. Hepatitis C screening tests are not required unless:

* Known history of HCV infection
* As mandated by local health authority

  * HIV-infected participants must have well-controlled HIV on antiretroviral treatment (ART), defined as:
* Participants on ART must have a CD4+ T-cell count ≥ 350 cells/mm^3 at the time of screening
* Participants on ART must have achieved and maintained virologic suppression defined as confirmed HIV ribonucleic acid (RNA) level below 50 or the LLOQ (below the limit of detection) using the locally available assay at the time of screening and for at least 12 weeks before screening
* It is advised that participants must not have had any AIDS-defining opportunistic infections within the past 12 months.
* Participants on ART must have been on a stable regimen, without changes in drugs or dose modification, for at least 4 weeks before study entry (day 1) and agree to continue ART throughout the study
* The combination ART regimen must not contain any antiretroviral medications that interact with CYP3A4 inhibitors/inducers/substrates (https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers)

  * Absolute neutrophil count (ANC) ≥ 1500/µL (collected within 10 days prior to the start of study)
  * Platelets ≥ 100 000/µL (collected within 10 days prior to the start of study)
  * Hemoglobin ≥ 9.0 g/dL or ≥ 5.6 mmol/L (collected within 10 days prior to the start of study). Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks
  * Creatinine ≤ 1.5 × upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) ≥ 30 mL/min for participant with creatinine levels > 1.5 × institutional ULN (collected within 10 days prior to the start of study)
* Creatinine clearance (CrCl) should be calculated per institutional standard

  * Total bilirubin ≤ 1.5 × ULN OR direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 × ULN (collected within 10 days prior to the start of study)
  * Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/ alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 × ULN (≤ 5 × ULN for participants with liver metastases) (collected within 10 days prior to the start of study)
  * International normalized ratio (INR) OR prothrombin time (PT) activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or activated partial thromboplastin time (aPTT) is within therapeutic range of intended use of anticoagulants (collected within 10 days prior to the start of study)

Exclusion Criteria:

* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137)
* Has received prior hysterectomy. (Prior lymphadenectomy permitted)
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks to /allocation
* Has received prior radiotherapy for cervical cancer
* Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded. Participants with low-risk early-stage prostate cancer (T1-T2a, Gleason score ≤ 6, and prostate specific antigen (PSA) < 10 ng/mL) either treated with definitive intent or untreated in active surveillance with stable disease are not excluded
* Has known active carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention
* Has severe hypersensitivity (≥ grade 3) to pembrolizumab and/or any of its excipients
* Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid)
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy
* History of Hepatitis B (defined as HBsAg reactive) or known active Hepatitis C virus (defined as detectable HCV RNA [qualitative]) infection.

Note: Testing for Hepatitis B or C is not required unless mandated by local health authority

* Has not adequately recovered from major surgery or has ongoing surgical complications
* Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment
* Has had an allogenic tissue/solid organ transplant
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2031-01-31 (Estimated); Study Completion 2032-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From the date of cycle 1 of chemotherapy (per protocol) to tumor progression or recurrence at any site, commencement of non-protocol anticancer therapy or death from any cause, whichever occurs first, up to 3 years
  Will be described using Kaplan-Meier plots and median estimates.
Incidence of adverse events | Up to 30 days after completion of study treatments

SECONDARY OUTCOMES:
PFS | From the date of cycle 1 of chemotherapy (per protocol) to tumor progression or recurrence at any site, commencement of non-protocol anticancer therapy or death from any cause, whichever occurs first, up to 3 years
  Will be described using Kaplan-Meier plots and median estimates.
Overall survival | Up to 3 years
  Will be described using Kaplan-Meier plots and median estimates.
Duration of response | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Dana M Chase, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (4):
- United States (4):
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - University of California San Diego (UCSD), San Diego, California
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Virginia Cancer Center, Charlottesville, Virginia